CLINICAL TRIAL: NCT03834155
Title: Enhancing Cardiac Rehabilitation Adherence Through Home-based Rehabilitation and Behavioral Nudges: ERA Nudge
Brief Title: Enhancing Cardiac Rehabilitation Through Behavioral Nudges
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-1290
Record Dates: First submitted 2018-12-20; First posted 2019-02-07 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Acute Myocardial Infarction; Percutaneous Coronary Intervention; Coronary Artery Disease; Valvular Disease; Chronic Stable Angina; Chronic Stable Heart Failure
MeSH Terms: conditions — Coronary Artery Disease; Angina, Stable

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hospital-based CR + Mobile Application (Experimental): Traditional hospital-based cardiac rehabilitation with mobile application.
  Interventions: Other: Hospital-based CR + Movn Application
- Choice CR + Mobile Application (Experimental): Choice of hospital or home-based cardiac rehabilitation with mobile application.
  Interventions: Other: Choice of Hospital or home-based CR + Movn Application
- Hospital-based CR + Mobile Application + Nudge (Experimental): Hospital-based cardiac rehabilitation with mobile application and nudges.
  Interventions: Other: Hospital-based CR + Movn Application + Nudge
- Choice CR + Mobile Application + Nudges (Experimental): Choice of Hospital or home-based cardiac rehabilitation with mobile application and nudges.
  Interventions: Other: Choice of Hospital or home-based CR + Movn Application + Nudge

INTERVENTIONS:
Other: Hospital-based CR + Movn Application — Participants will be randomly assigned to a group that will receive hospital-based CR and access to the Movn mobile application.
  Arms: Hospital-based CR + Mobile Application
Other: Choice of Hospital or home-based CR + Movn Application — Participants will be randomly assigned to a group that has opportunity to opt in to hospital-based cardiovascular rehabilitation or home-based cardiovascular rehabilitation. All will have access to the Movn Application.
  Arms: Choice CR + Mobile Application
Other: Hospital-based CR + Movn Application + Nudge — Participants will be randomly assigned to a group that will receive hospital-based CR and access to the Movn mobile application, plus encouraging nudge messages.
  Arms: Hospital-based CR + Mobile Application + Nudge
Other: Choice of Hospital or home-based CR + Movn Application + Nudge — Participants will be randomly assigned to a group that has opportunity to opt in to hospital-based cardiovascular rehabilitation or home-based cardiovascular rehabilitation. All will have access to the Movn Application, plus encouraging nudge messages.
  Arms: Choice CR + Mobile Application + Nudges

SUMMARY:
Adherence to cardiac rehabilitation is poor, and worse for minorities, women, and those with lower levels of education. Patients less likely to be referred to and complete cardiac rehab are at highest risk of adverse outcomes and thus have the most to gain from participation in cardiac rehab. To improve participation, healthcare systems need to limit barriers to enrollment and promote adherence to rehabilitation.

DETAILED DESCRIPTION:
This study aims to (1) iteratively develop and program a theoretically informed technology-based nudge message library for a diverse patient population using multiple and iterative N of 1 within subject studies. Investigators will also engage patient, provider and health systems stakeholders in designing and refining the messages. (2)Develop a one-page decision aid tool to present information designed with principles of shared decision making including pros and cons of hospital and home-based rehabilitation. Investigators will engage patients, providers, and health systems stakeholders to provide feedback on the information sheet. (3) Conduct a 2x2 factorial design randomized trial of a) choice and b) nudge messaging to improve primary outcome of CR adherence. Secondary outcomes will include enrollment and completion of CR, exercise capacity, patient engagement, quality of life, hospitalizations, and healthcare utilization. The study will additionally evaluate the interventions using a mixed methods approach applying the RE-AIM (reach, effectiveness, adoption, implementation, and maintenance) framework and a cost-effectiveness analysis. The cost-effectiveness analysis sub-study will evaluate the implementation cost of home-based and hospital-based cardiac rehabilitation programs in addition to the incremental cost effectiveness ratios for each intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myocardial infarction, percutaneous coronary intervention, coronary artery bypass graft, valvular heart surgery, chronic stable angina, and/or chronic stable heart failure with left ventricular systolic dysfunction.
* 18 year of age or older
* Access to a cell phone with text messaging capability
* English or Spanish speaking

Exclusion Criteria:

* Medical director's decision based on high-risk assessment
* Enrolled in hospice or palliative care
* Being intoxicated or otherwise unable to consent to participate

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2019-05-17 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Adherence to cardiovascular rehabilitation measured by self-report in the Movn Application or through EHR/exercise physiologist report in RedCap | 12 weeks
  Attendance for 4 weeks (8 or more) exercise sessions for hospital-based CR or logging exercise data for 4 weeks for home-based rehabilitation.

SECONDARY OUTCOMES:
Active enrollment of 280 DH participants | 3.5 yrs
  Attending one visit following baseline visit or logging exercise data at least once for home-based CR.
Completion of cardiovascular rehabilitation as defined by attending or logging 18 exercise sessions | 12 weeks
  Attending or logging 18 exercise sessions
Exercise capacity measured by a 6-minute walk test. | 12 weeks
  Exercise capacity will be measured at the index visit, 6 weeks, 12 weeks.
Patient activation and engagement will be measured using the 13-item Patient Activation Measure (PAM) | 12 weeks
  The low-literacy version of the 13-item Patient Activation Measure (PAM), both in English and Spanish, will be used to assess the effect of the intervention on patient activation. This validated and predictive tool assesses patient knowledge, skill and confidence in self-management. A single point change in PAM score is clinically meaningful and increases in the PAM are associated with increased self-management behavior. The PAM will be measured at the index visit, 6 weeks, 12 weeks.
Reported quality of life measured by Ferrans and Powers Quality of Life Index | 12 weeks
  The Ferrans and Powers Quality of Life Index (QLI) will be used to assess quality of life. The QLI is a 35 question instrument that uses a 6 point scale ranging from "very unimportant (lower end of the scale)" to "very important (higher end of the scale)". The outcomes of these scales are averaged to compute the total score. The QLI is valid, reliable, sensitive to change in both CR and PR populations, and is available in English and in Spanish. The QLI will be administered at the index visit, 6 weeks and 12 weeks.
Number of participants hospitalized over four months using EHR review and ICD-10s | 6 months
  All-cause hospitalizations will be ascertained via the EHR using ICD-10 codes. Follow-up for hospitalizations will occur through 6 months.
Number of participants who attend or log of 36 cardiovascular rehabilitation sessions measured by self-report in the Movn Application or through EHR/exercise physiologist report in RedCap | 12 weeks
  Attending or logging 36 exercise sessions.
Type of healthcare utilization by individual participants, defined by routine clinical visits. Urgent care and emergency department visits will be measured using EHR. | 6 months
  Healthcare utilization, defined by routine clinical visits. Urgent care and emergency department visits will be measured using EHR.
Safety measures to track injury from exercise will be assessed using EHR | 12 weeks
  Injury from exercise will be assessed using EHR including hospitalizations, emergency department visits, urgent care visits and mortality safety endpoints.
  They will be captured at the time of occurrence and records will be reviewed by the DSMB.
Socioeconomic and clinical data will be collected from EHR. | 3.5 yrs
  Sociodemographic and clinical data will be collected from DH registration files including age, gender, self-reported race/ethnicity, primary language preference, comorbid diagnoses (hypertension, diabetes, chronic kidney disease, depression, substance abuse), measures of disease severity (left ventricular ejection fraction, FEV1) and medications.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Peterson, MD, MSPH, Principal Investigator — Denver Health and Hospital Authority
Locations (1):
- Denver Health and Hospital Authority, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gupta P, Fletcher DR, Durfee J, Martinez M, Hajoglou A, Waughtal J, Bull S, Peterson PN. Enhancing cardiac rehabilitation adherence through home-based rehabilitation and behavioral nudges: The ERA nudge study design and rationale. Am Heart J. 2025 Dec;290:17-28. doi: 10.1016/j.ahj.2025.05.010. Epub 2025 May 16. PMID 40383506